CLINICAL TRIAL: NCT04639700
Title: A Pilot Study to Evaluate the Feasibility of an Intervention for Caregivers of Patients Who Have Recently Undergone HSCT
Brief Title: Intervention for Caregivers of Patients Who Have Recently Undergone HSCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE14Z20
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Caregiver Anxiety; Caregiver Distress; Caregiver Health Related QOL
Keywords: Hematopoietic stem cell transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psycho-educational intervention (Experimental): All participants will receive receive 4 individual sessions with an interventionist in addition to the standard post-hospital HSCT information for patient follow-up care as provided by the patient's oncologist
  Interventions: Behavioral: Psycho-educational intervention

INTERVENTIONS:
Behavioral: Psycho-educational intervention — Participant will be sent a baseline survey, and will then be contacted by the interventionist to complete 4 sessions, which feature the following areas:
  Session 1: Identifying CG Needs for Information & Support, Communication with Healthcare Team
  Session 2: Communication with Patient and Family
  Session 3: Self-care: Emotional & Spiritual Needs, Self-care: Physical Needs
  Session 4: Re-Assessing Needs, Planning for the future

SUMMARY:
The purpose of this study is to find out if providing support to caregivers of patients who have recently had a HSCT is possible and helpful.

DETAILED DESCRIPTION:
This study will test the feasibility, acceptability, usability, satisfaction and preliminary efficacy of a behavioral (psychoeducation) intervention. All participants will receive the standard post-hospital HSCT information for patient follow-up care as provided by the patient's oncologist. In addition, the all participants will receive 4 individual sessions with an interventionist.

ELIGIBILITY:
Inclusion Criteria:

* An adult family or friend of a patient who has been discharged from the hospital in the past 1-2 weeks after receiving HSCT
* Identifies himself/herself as the caregiver who will be responsible for the patient's care post-HSCT
* Has English as their primary language

Exclusion Criteria:

-Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Acceptability Scale scores | At 2 months
  Caregiver Acceptability as measured by Acceptability Scale scores. Overall score ranging from 6-30. According to prior research, a score of 80% of higher (total score of 24 or higher) is considered acceptable for use.
System Usability Scale scores | At 2 months
  Caregiver Usability as measured by the System Usability Scale. This is a 10 item scale scored on a 5 point Likert scale with total summed scores ranging from 0-50. Total scores are multiplied by 2 to produce an overall score ranging from 0-100 with scores > 68 considered to be above average usability
Mean caregiver satisfaction scores | At the end of each intervention session and end of study evaluation, up to 2 months
  Caregiver Satisfaction scores as measured by Likert Scale. After completing each module, they will be sent via REDCap a single item evaluation scale (0 -10; 0=Not at all satisfied; 10=Highly satisfied). Scores >7 will be considered acceptable. Mean and standard deviation will be reported.
Percent of enrollment of eligible participants | At 2 months
  Feasibility as measured by percent of enrollment of eligible participants
Percent of participants completing intervention | At 2 months
  Feasibility as measured by intervention completion
Retention rate | At 2 months
  Feasibility as measured by percent of participants retained in full study (aim: 90% retention at the end of the 2-month intervention)
Average time to recruit dyads in months | At 2 months
  Feasibility as measured by time to identify and recruit dyads in months (benchmark 3 months)
Data collection completion rate | At 2 months
  Feasibility as measured by completion of data collection across study timepoints

SECONDARY OUTCOMES:
NCCN Distress Thermometer scores | At baseline and at 2 months
  Caregiver Distress as measured by NCCN Distress Thermometer scores
PROMISR Short Form v1.0 - Anxiety | At baseline and at 2 months
  Caregiver Anxiety as measured by PROMISR Short Form v1.0 - Anxiety scores. Scores range from 1 to 5, with higher scores indicating worse anxiety
PROMISRv.1.2 - GlobalHealth scores | At baseline and at 2 months
  Caregiver Health Related Quality of Life as measured by PROMISRv.1.2-GlobalHealth scores. HRQOL scores range from 1 to 5, with higher scores indicating better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sara Douglas, PhD, RN, Principal Investigator — Case Western Reserve University

IPD SHARING:
Plan to Share IPD: No
This is a pilot study to only test the intervention so the data would not be useful to participants until a larger study (with control and intervention groups) is completed in the future